CLINICAL TRIAL: NCT06434727
Title: A Retrospective Multicenter Study for Intuitive 3D Models (I3DM), During Simulated Preoperative Surgical Planning for Anatomic Lung Resection and Lower Anterior Resection Procedures
Brief Title: Evaluating Intuitive 3D Models in Preoperative Surgical Planning for Thoracic and Colorectal Procedures.
Acronym: ISI-I3DM-01
Status: Recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-I3DM-01
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2024-10

CONDITIONS: Thoracic; Colorectal Disorders
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thoracic Group: Anatomic Lung Resection (Segmentectomy or Lobectomy) Procedures
  Interventions: Other: observational study
- Colorectal Group: Lower Anterior Resection Procedures
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Observational Study

SUMMARY:
The Study Objective: To evaluate the clinical utility of a 3D model with 2D CT/MRI scans during simulated preoperative surgical planning of open, laparoscopic, or robotic-assisted anatomic lung resection (segmentectomy, lobectomy) or Lower Anterior Resection (LAR) procedures.

DETAILED DESCRIPTION:
This is a Retrospective study evaluating the clinical utility of a 3D model with 2D CT/MRI scans during simulated preoperative surgical planning of open, laparoscopic, or robotic-assisted anatomic lung resection (segmentectomy, lobectomy) or Lower Anterior Resection (LAR) procedures.

ELIGIBILITY:
Inclusion Criteria:

- DICOM images from Subjects 18 years or older who have undergone either anatomic lung resection (segmentectomy, lobectomy) or a Lower Anterior Resection procedure

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years or older who have undergone either anatomic lung resection (segmentectomy, lobectomy) or a Lower Anterior Resection procedure will be considered for this study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Utility of 3D Model vs standard 2D in Preoperative Surgcial Planning | 2 months
  Surgeon questionnaires evaluating their preoperative surgical plan

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - The Feinstein Institutes for Medical Research, Manhasset, New York
  - The Ohio State University, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No